CLINICAL TRIAL: NCT04272957
Title: A Phase I, Open-Label, Multicenter Study to Assess the Safety, Pharmacokinetics and Efficacy of HMPL-306 in Patients of Relapsed/Refractory Myeloid Leukemia/Neoplasms With IDH1 and/or IDH2 Mutation
Brief Title: A Study of HMPL-306 in Patients With IDH1 and/or IDH2 Mutation of Relapsed/Refractory Myeloid Leukemia/Neoplasms
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-306-00CH1
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: HMPL-306; IDH1 Mutation; IDH2 Mutation; Acute myeloid leukemia; Myelodysplastic symdrome; Chronic myelomonocytic leukemia; Myeloid Leukemia/Neoplasms
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-306 (Experimental): HMPL-306 administered continuously as a single agent orally every day in a 28-day cycle.
  Interventions: Drug: HMPL-306

INTERVENTIONS:
Drug: HMPL-306 — HMPL-306 administered continuously as a single agent starting at 25 mg orally every day in a 28-day cycle and dose escalation is planned up to 200mg. Subjects may continue treatment with HMPL-306 until disease progression, development of other unacceptable toxicity or hematopoietic stem cell transplant.

SUMMARY:
Phase I, multicenter study to evaluate the safety, pharmacokinetics, pharmacodynamics and efficacy of HMPL-306 in Patients of Relapsed/Refractory Myeloid Leukemia/Neoplasms with IDH1 and/or IDH2 Mutation.

DETAILED DESCRIPTION:
The purpose of this Phase I, multicenter study is to evaluate the safety, pharmacokinetics, pharmacodynamics and efficacy of HMPL-306 in Patients of Relapsed/Refractory Myeloid Leukemia/Neoplasms with IDH1 and/or IDH2 Mutation. The first stage of the study is a dose escalation phase where cohorts of patients will receive ascending oral doses of HMPL-306 to determine maximum tolerated dose (MTD) and/or the recommended Phase II dose. The second stage of the study is a dose expansion phase where three cohorts of patients will receive HMPL-306 to further evaluate the safety, tolerability, and clinical activity of the recommended Phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* Signed Informed Consent Form;
* Relapsed/refractory Acute myeloid leukemia (AML), myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia(CMML) and others myeloid neoplasm;
* IDH1 and/or IDH2 mutated disease status as assessed by local laboratory;
* Cooperative Oncology Group (ECOG) performance status of 0-2;
* Subjects must be amenable to serial bone marrow biopsies, peripheral blood sampling, and urine sampling during the study.

Exclusion Criteria:

* Previously treated with any prior IDH1 inhibitor, IDH2 inhibitor, or IDH1/IDH2 double-targeted therapy and had disease progression during treatment;
* with known involvement or clinical symptoms of central nervous system (CNS);
* Patients who have undergone HSCT within 60 days;
* Without adequate liver or kidney function;
* With known infection with active hepatitis B or C;
* With known infection with human immunodeficiency virus (HIV);
* History of clinically significant or active cardiac disease;
* Active clinically significant infection;
* Taking known strong cytochrome P450 (CYP) 2C8 inducers or inhibitors;
* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Incidence of adverse events | Baseline up to the last patient has completed the 24 weeks of treatment
  Incidence of adverse events.
Maximum tolerated dosage (MTD) and/or recommended phase 2 dosage (RP2D) | Baseline up to the last patient has completed the 24 weeks of treatment
  Measured by adverse event profile.

SECONDARY OUTCOMES:
Cmax (Cycle 1 Day 1) of HMPL-306 | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11, 24, 48, 72, 120 and 168 hours after start
  Cmax: maximum observed drug concentration in measured matrix after single dose administration.
AUC(0-24) (Cycle 1 Day 1) of HMPL-306 | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11, 24, 48, 72, 120 and 168 hours after start
  AUC: area under the concentration vs. time curve from zero to infinity after single (first) dose.
AUC(0-tlast) (Cycle 1 Day 1) of HMPL-306 | Pre-dose, 10 minutes, 1, 1.5, 2, 3, 5, 8, 11, 24, 48, 72, 120 and 168 hours after start
  AUC from time zero to the last data point.
Objective Response Rate (ORR) | Baseline up to the last patient has completed the 24 weeks of treatment
  proportion of patients with confirmed complete response (CR) and partial response (PR).
Duration of response (DOR) | Baseline up to the last patient has completed the 24 weeks of treatment
  DOR is defined as the time from the date of first observed tumor response (Complete response (CR) or Partial response (PR)) until first subsequent disease progression or until death (if death occurs before progression is documented) due to any cause.
Progression-free survival (PFS) | Baseline up to the last patient has completed the 24 weeks of treatment
  PFS is defined as the time from enrollment (i.e., date of treatment assignment) to disease progression.
Overall survival (OS) | Baseline up to the last patient has completed the 24 weeks of treatment
  OS is defined as the time from enrollment (i.e., date of treatment assignment) until death from any cause or until the last date the patient is known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Weiss Yang, Study Director — Hutchison MediPharma Ltd
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu L, Wei X, Zhao W, Hu Y, Li J, Dong Y, Gong T, Zhang X, Xu Y, Zhang Y, Xu C, Zhang C, Cai Z, Jing H, Mi R, Wu W, He W, Wang H, Tang Q, Jiang Z, Liu H, Chen G, Sun J, Chen J, Yan S, Yan H, Wangwu J, Zhong Z, Wang L, Fan S, Shi M, Su W, Huang X. HMPL-306 in relapsed or refractory IDH1- and/or IDH2-mutated acute myeloid leukemia: A phase 1 study. Med. 2025 Jun 13;6(6):100575. doi: 10.1016/j.medj.2025.100575. Epub 2025 Jan 31. PMID 39892383